CLINICAL TRIAL: NCT01413789
Title: Measurement and Comparison of the Occlusive and Hydrating Capacity of Three Silicone Gels: BAP Scar Gel, Dermatix, Kelocote and One Gel- Cream: Alhydran
Brief Title: Measurement and Comparison of the Occlusive and Hydrating Capacity of Three Silicone Gels and One Gel Cream
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/350
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Scar Tissue or Healthy Skin
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients and healthy volunteers (Experimental): Patients with healed full thickness burns and healthy volunteers will be included in the study
  Interventions: Drug: Dermatix; Drug: Kelocote; Drug: BAP scar gel; Drug: Alhydran; Drug: Bap Scar Care T; Drug: Bap Scar Care S; Drug: Mepiform; Drug: Scar Ban Elastic

INTERVENTIONS:
Drug: Dermatix — 1 application of Dermatix
Drug: Kelocote — 1 application of Kelocote
Drug: BAP scar gel — 1 application of BAP scar gel
Drug: Alhydran — 1 application of Alhydran
Drug: Bap Scar Care T — 1 application of BAP Scar Care T
Drug: Bap Scar Care S — 1 Application of Bap Scar Care S
Drug: Mepiform — 1 application of Mepiform
Drug: Scar Ban Elastic — 1 application of Scar Ban Elastic

SUMMARY:
Study hypothesis: Is Alhydran gel-cream as efficient as silicone gel for skin occlusion and hydration?

For this study 16 volunteers and ten patients with healed full thickness burns will be included.

After a short period of acclimatization four test areas will be determined. For healthy volunteers the standard zones are located on the inner forearm, two on each forearm.

For patients with healed burns the 4 test zones are located on either the healed donor site or the healed skin grafted area.

In each test zone baseline measurements will be taken before application of the products.After application of the three silicone gels and the hydrating gel cream the trans epidermal water loss (TEWL) and the moisture content of the stratum corneum will be measured by using the TEWAmeter®TM300 and the Corneometer® CM825 (Courage & Khazaka).

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers or patients with healed full thickness burns and donor sites
* not pregnant
* age>18 years
* male or female
* written authorisation of the patient or volunteer is required.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The occlusive and hydrating capacity of the products. | 1 hour after application
  Measurements will be done by using the TEWAmeter® for measurement of the Trans Epidermal Waterloss and the Corneometer® 825CM for measurement of the moisture content of the stratum corneum (Courage & Khazaka). For this study no risk factors are determined.

SECONDARY OUTCOMES:
The occlusive and hydrating capacity of the products. | 2 hours after application
  Measurements will be done by using the TEWAmeter® for measurement of the Trans Epidermal Waterloss and the Corneometer® 825CM for measurement of the moisture content of the stratum corneum (Courage & Khazaka). For this study no risk factors are determined.
The occlusive and hydrating capacity of the products. | 3 hours after application
  Measurements will be done by using the TEWAmeter® for measurement of the Trans Epidermal Waterloss and the Corneometer® 825CM for measurement of the moisture content of the stratum corneum (Courage & Khazaka). For this study no risk factors are determined.

CONTACTS AND LOCATIONS:
Overall Officials: S. Monstrey, MD PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be